CLINICAL TRIAL: NCT01552603
Title: Sensor-controlled Insulin- and Glucagon Delivery in Subjects With Type 1 Diabetes: Testing of an Automated System in a Supervised Inpatient Setting
Brief Title: Artificial Pancreas Control System in an Inpatient Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Legacy Health System (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, W. Kenneth Ward, Senior Scientist, Legacy Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011.11
Record Dates: First submitted 2012-02-22; First posted 2012-03-13 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-04

CONDITIONS: Type I Diabetes Mellitus
Keywords: glucose sensors; artificial pancreas; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Artificial Pancreas Control (Experimental): Type 1 Diabetes Mellitus subjects who fit the inclusion/exclusion criteria will undergo artificial pancreas closed-loop study for 28 hours. For the entire study, the adaptive component of Artificial Pancreas Control Software will be used to control the subject's blood glucose.
  Interventions: Device: Artificial Pancreas Control Software

INTERVENTIONS:
Device: Artificial Pancreas Control Software — This master controller software is used in conjunction with two subcutaneous continuous glucose monitoring systems and two Omnipod pumps, one for administering aspart insulin (NovoLog) and one for administering glucagon (GlucaGen), to control blood glucose levels. The insulin and glucagon infusion rates are determined by an automated version of the Adaptive Proportional Derivative (APD) insulin and glucagon control algorithm.

SUMMARY:
The purpose of this study is to verify an automated system of blood glucose control in Type I Diabetics. The automated system consists of the investigational Artificial Pancreas Control software (APC), two blood glucose sensors, and two hormone pumps, one for delivering insulin to lower blood sugar, and the second for delivering glucagon to raise blood sugar. The blood glucose sensors relays information to the Artificial Pancreas software, which uses the Adaptive Proportional Device algorithm to determine the rate of insulin and glucagon infusion by the hormone pumps. In prior studies, the Adaptive Proportional Device algorithm has been verified, but required manual input into the computer and hormone pumps. This study differs in that it uses a fully automated system under the control of the Artificial Pancreas Control software. The importance of this change is that it is the next step to enable outpatient use of automated, closed loop blood glucose control.

DETAILED DESCRIPTION:
The objective of the current human study is to verify the components of the Artificial Pancreas Control system during an inpatient study. This master controller software is designed to be used in conjunction with two subcutaneous continuous glucose monitoring systems to regulate blood glucose levels as well as two Omnipod pumps, one for administering insulin and one for administering glucagon. The sensors communicate wirelessly with two sensor receivers which will be interfaced with the APC by wireless USB connection. The insulin and glucagon pumps will be controlled by the APC through a wireless USB connection. The algorithm included in the APC is an automated version of the Adaptive Proportional Derivative (APD) insulin and glucagon control algorithm, which was previously studied as an investigational device. The APD has been studied in vivo (in 28 experiments, each 33 hr in length, with manual adjustment of pumps) and no serious adverse effects were noted. Manual input of the glucose sensor data and insulin/glucagon infusion rates will no longer be necessary. The APC will be tested in vivo during 28 hour experiments in an inpatient setting in preparation for outpatient testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes mellitus for at least 1 year.
* Male or female subjects 21 to 65 years of age.
* Current use of an insulin pump.
* Willingness to follow all study procedures, including attending all clinic visits.
* Willingness to sign informed consent and HIPAA documents.

Exclusion Criteria:

* Pregnancy or Lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 1 month after participating in the study. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
* Renal insufficiency (serum creatinine of 2.0 mg/dL or greater).
* Serum ALT or AST equal to or greater than 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as a serum albumin of less than 3.3 g/dL; or serum bilirubin of over 2.
* Adrenal insufficiency
* Hematocrit of less than or equal to 34%.
* A history of cerebrovascular disease or coronary artery disease regardless of the time since occurrence.
* Congestive heart failure, NYHA class III or IV.
* Diagnosis of 2nd or 3rd degree heart block or any arrhythmia judged by the investigator to be exclusionary.
* Any active infection.
* Visual impairment preventing reading of glucose meter values or continuous glucose monitoring device.
* Physical impairment impeding the ability to use a glucose meter or glucose monitoring device.
* Active foot ulceration.
* Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
* Active alcohol abuse, substance abuse, or severe mental illness (as judged by the principal investigator).
* Active malignancy, except basal cell or squamous cell skin cancers.
* Major surgical operation within 30 days prior to screening.
* Seizure disorder.
* Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
* Current administration of oral or parenteral corticosteroids.
* Use of an investigational drug within 30 days prior to screening.
* Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
* Allergy to aspart insulin.
* Allergy to glucagon.
* Past history of pheochromocytoma or a family history of MEN 2, neurofibromatosis, or von Hippel-Lindau disease.
* Insulin resistance requiring more than 200 units per day.
* Need for uninterrupted treatment of acetaminophen.
* Intolerance of mild hypoglycemia (glucose 60-70 mg/dl).
* History of hypoglycemic unawareness.
* Insulin antibody level of ≥ 100 µUnits/ml.
* C peptide level of ≥0.5 ng/ml.
* Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen.
* Any reason the principal investigator deems exclusionary

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W K Ward, MD, Principal Investigator — Legacy Health Research
Locations (2):
- United States (2):
  - Legacy Good Samaritan Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon

REFERENCES:
- [Background] El Youssef J, Castle JR, Branigan DL, Massoud RG, Breen ME, Jacobs PG, Bequette BW, Ward WK. A controlled study of the effectiveness of an adaptive closed-loop algorithm to minimize corticosteroid-induced stress hyperglycemia in type 1 diabetes. J Diabetes Sci Technol. 2011 Nov 1;5(6):1312-26. doi: 10.1177/193229681100500602. PMID 22226248

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Artificial Pancreas Control
Started | 14
Completed | 13
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Artificial Pancreas Control
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent of Time in Target Blood Glucose Range
Description: Mean percent of time venous blood glucose was sampled between 70-180 mg/dl
Time Frame: all 28 hour studies
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Artificial Pancreas Control
Number analyzed (Participants) | 13
percentage of time | 62.4 (7.0)

2. Secondary Outcome: Mean Deviation From Target Blood Glucose
Description: Mean difference of venous blood glucose from glucose target. Daytime venous blood glucose values (7am-11pm) subtracted from daytime target of 115 mg/dl. Nighttime venous blood glucose values (11pm-7am) subtracted from nighttime target of 140 mg/dl. This is a metric of how successful the closed loop algorithm was at controlling glucose.
Time Frame: all 28 hour studies
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Artificial Pancreas Control
Number analyzed (Participants) | 13
mg/dl | 59.9 (51.6)

ADVERSE EVENTS:
Arm/Group | Artificial Pancreas Control
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Artificial Pancreas Control (N=14)
hematoma (Blood and lymphatic system disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes